CLINICAL TRIAL: NCT07369219
Title: Investigating the Effect of a Care Intervention Implemented in Stoma Patients Receiving Care Based on Enhanced Recovery Propositions on Patient Outcomes and Home Care Management: A Mixed Methods Study
Brief Title: Effect of a Nursing Care Intervention on Outcomes of Stoma Patients Within an Enhanced Recovery Framework
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Özlem Kıvanç, PhD student, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Approval number 2025-03/147
Record Dates: First submitted 2025-05-16; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Home Care; Stoma; Enhanced Recovery
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Routine hospital discharge education, usual stoma care follow-up, and standard postoperative monitoring without the additional structured education booklet or planned telephone follow-up.
  Interventions: Other: Standard maintenance therapy
- intervention group (Experimental): A structured discharge education program supported with a home-care booklet and scheduled telephone follow-up at postoperative days 3, 7, 10, and 30.
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Educational intervention — A structured discharge education program supported with a home-care booklet and scheduled telephone follow-up at postoperative days 3, 7, 10, and 30.
  Arms: intervention group
Other: Standard maintenance therapy — Routine postoperative stoma care and standard hospital discharge education provided according to institutional protocols. Usual care includes routine monitoring of the stoma site, general postoperative recovery assessment, complication screening, and standard follow-up visits without the structured education booklet or scheduled telephone follow-up program.
  Arms: Control Group

SUMMARY:
Colorectal cancer is one of the most common cancers in the world and affects a large number of people every year. Surgical intervention and neoadjuvant treatment are mostly preferred for treatment, and temporary or permanent stoma is often opened. Complications that are difficult to manage may arise due to the treatment itself, the disease or the stoma. Complications that are difficult to manage carry a high risk of re-hospitalization. Patients receive limited support during the transition from hospital to home and at home. Patients and their relatives are often alone in home care management until the routine check-up process. Especially patients who are not well prepared for discharge and inadequate in stoma management may not know how to apply care practices during this period at home and the situations they should pay attention to in case of complications. Conditions that can be managed well in the hospital may get out of control when the patient goes home and may cause unplanned re-admissions to the hospital if there is not enough follow-up. Inadequate patient follow-up after surgery may cause patients to be anxious and therefore may cause re-hospitalization due to the inability to manage the home care process in a controlled manner.

Although it is known that the duration of hospital stay is shortened with advanced improvement suggestions, different results are remarkable in studies on hospital readmissions, reoperations, developing complications and survival. Since the care needs of patients after surgical intervention vary, there is a need for individualized and evidence-supported suggestions. Currently, advanced improvement suggestions do not include the answer to the question and roadmap of how patients will be followed at home after discharge. The surgical journey should be followed with comprehensive care application steps that are a continuation of evidence-based practices that start from the moment the patient is admitted to the hospital, making them feel that they are not alone during the recovery process they will spend at home after being discharged. The provision of home care management is important for the continuity of the recovery process. Although there are various application models used in the literature for the purpose of preparing and following up on the discharge process, no study has been found that focuses on comprehensive discharge preparation and home care management of stoma patients receiving care in line with advanced recovery recommendations. In this sense, it is believed that the study will be a fundamental study in terms of developing a fourth phase, post-discharge home care management, which is the continuation of the pre-, intra- and post-operative process as included in advanced recovery guidelines and a gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study

  * Be 18 years of age or older
  * Be able to communicate in Turkish
  * Have no visual or hearing impairment
  * Elective colorectal surgery in line with advanced treatment recommendations Having a stoma opened for the first time due to colorectal cancer

Exclusion Criteria:

* patients who did not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
KATZ Activities of Daily Living (ADL) Scale | Baseline (pre-discharge) and postoperative day 30
  If the individual can do their ADL independently, they are given 3 points, if they are partially assisted, they are given 2 points, if they cannot do it at all, they are given 1 point and the evaluation is made accordingly. In the evaluation made according to this scale, 0-6 points are evaluated as dependent, 7-12 points as partially dependent, and 13-18 points as independent. Accordingly, as the score obtained from the scale increases, dependency decreases.
EORTC QLQ-C30 Quality of Life Scale | Baseline (pre-discharge) and postoperative day 30
  The lowest total score that patients can get from the functional score, symptom score and general health score is 0, and the highest score is 100. A high score from the functional scales indicates a healthy functional level, a high score from the general health status scale indicates a high quality of life, and a high score from the symptom scale indicates that symptoms are experienced intensely and the level of the problem is high.
Stoma-Self-Efficacy Scale | Baseline (pre-discharge) and postoperative day 30
  The total score of the scale ranges from 22 to 110, with higher scores indicating increased self-efficacy levels of patients.
Readiness for Discharge Scale | Up to 30 days after the patient's hospitalization date.
  If the scale dimensions score was ≥7, the patient was considered ready for discharge, and if it was <7, it was considered not ready.

SECONDARY OUTCOMES:
Day of hospital stay | Up to 30 days after the patient's hospitalization date.
complications | Up to postoperative day 30
Readmisson | Within 30 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Maslak Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data is patient specific, therefore, other data will not be shared except for the research results.

REFERENCES:
- [Result] Storm M, Morken IM, Austin RC, Nordfonn O, Wathne HB, Urstad KH, Karlsen B, Dalen I, Gjeilo KH, Richardson A, Elwyn G, Bru E, Soreide JA, Korner H, Mo R, Stromberg A, Luras H, Husebo AML. Evaluation of the nurse-assisted eHealth intervention 'eHealth@Hospital-2-Home' on self-care by patients with heart failure and colorectal cancer post-hospital discharge: protocol for a randomised controlled trial. BMC Health Serv Res. 2024 Jan 4;24(1):18. doi: 10.1186/s12913-023-10508-5. PMID 38178097
- [Result] Lin L, Fang Y, Wei Y, Huang F, Zheng J, Xiao H. The effects of a nurse-led discharge planning on the health outcomes of colorectal cancer patients with stomas: A randomized controlled trial. Int J Nurs Stud. 2024 Jul;155:104769. doi: 10.1016/j.ijnurstu.2024.104769. Epub 2024 Apr 5. PMID 38676992
- [Result] van Rooijen S, Carli F, Dalton S, Thomas G, Bojesen R, Le Guen M, Barizien N, Awasthi R, Minnella E, Beijer S, Martinez-Palli G, van Lieshout R, Gogenur I, Feo C, Johansen C, Scheede-Bergdahl C, Roumen R, Schep G, Slooter G. Multimodal prehabilitation in colorectal cancer patients to improve functional capacity and reduce postoperative complications: the first international randomized controlled trial for multimodal prehabilitation. BMC Cancer. 2019 Jan 22;19(1):98. doi: 10.1186/s12885-018-5232-6. PMID 30670009
- [Result] Li MZ, Wu WH, Li L, Zhou XF, Zhu HL, Li JF, He YL. Is ERAS effective and safe in laparoscopic gastrectomy for gastric carcinoma? A meta-analysis. World J Surg Oncol. 2018 Jan 26;16(1):17. doi: 10.1186/s12957-018-1309-6. PMID 29373978
- [Result] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435